CLINICAL TRIAL: NCT02818218
Title: Superior Vena Cava (SVC) Diameter and Collapsibility Index and Its Relationship to Central Venous Pressure (CVP) Measurements in Patients Undergoing Liver Transplantation
Brief Title: Superior Vena Cava and Its Relationship to Central Venous Pressure Measurements in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 16-307
Record Dates: First submitted 2016-04-11; First posted 2016-06-29 (Estimated); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Liver Transplant — liver transplant recipient surgery

SUMMARY:
Consecutive patients undergoing liver transplant surgery will be included in the study. Before surgical incision, during the preanhepatic phase, during the anhepatic phase, during the postanhepatic phase and following closure of the deep fascial layer of the anterior abdominal wall simultaneous measurement of SVC diameter, SBC collapsibility index and CVP will be recorded.

DETAILED DESCRIPTION:
Central venous pressure (CVP) measured invasively through a central venous catheter in the internal jugular vein or through a right atrial port of a pulmonary artery catheter is commonly used during liver transplant surgery. CVP measurements at the SVC-RA junction are a function of circulating blood volume, right ventricle function, intrathoracic pressure. CVP measurements can also be affected by the presence of tricuspid regurgitation. Because central venous pressure measurements are determined by several factors and do not predict the response to subsequent fluid bolus administration, they are considered "static measures" and are poor indicators of fluid responsiveness.

Given the entirely intrathoracic location of the superior vena cava (SVC), its diameter and collapsibility with positive pressure ventilation it is a potentially attractive method of non-invasively estimating CVP.

SVC diameter and collapsibility index, dynamic measures of fluid responsiveness have been successfully utilized as echocardiographic indices for fluid responsiveness in ventilated septic patients. Whether SVC collapsibility is correlated with CVP measurements in liver transplant patients is not known.

Consecutive patients undergoing liver transplant surgery will be included in the study. Before surgical incision, during the preanhepatic phase, during the anhepatic phase, during the postanhepatic phase and following closure of the deep fascial layer of the anterior abdominal wall simultaneous measurement of SVC diameter, SBC collapsibility index and CVP will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* undergoing liver transplantation surgery (cadaveric and living related)

Exclusion Criteria:

* Contraindication to Transesophageal echocardiography

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing liver transplantation surgery (cadaveric and living related)
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, Principal Investigator — Outcomes Research Institute
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Liver Transplantation Patients: We conducted a prospective, single-group, observational study in order to assess the correlation between the diameter of the superior vena cava (SVC) and the central venous pressure (CVP) in patients undergoing liver transplantation surgeries. Aside for the transthoracic echocardiogram necessary to measure the SVC, no additional treatments were applied to the patient population.
Period: Overall Study
Arm/Group | Liver Transplantation Patients
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Liver Transplantation Patients
Number analyzed (Participants) | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [55 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48
  Other | 10
Current smoker [Count of Participants; unit: Participants] | 26
BMI [Mean (Standard Deviation); unit: kg/m2] | 29 (6)
ASA (American Society of Anesthesiologists) physical status [Count of Participants; unit: Participants]
  3 (Severe systemic illness) | 3
  4 (Life-threatening systemic illness) | 53
  5 (Not expected to survive without the operation) | 2
Alcoholic Cirrhosis [Count of Participants; unit: Participants] | 18
Primary Billary Cirrhosis [Count of Participants; unit: Participants] | 1
Hepatocellular Carcinoma [Count of Participants; unit: Participants] | 17
Primary Sclerosing Cholangitis [Count of Participants; unit: Participants] | 7
Non-alcoholic Steatohepatosis (NASH) [Count of Participants; unit: Participants] | 39
Viral Cirrhosis [Count of Participants; unit: Participants] | 16

OUTCOME MEASURES:

1. Primary Outcome: Central Venous Pressure (CVP)
Description: Central Venous Pressure (CVP) reflects the amount of blood returning to the heart (venous return) and the ability of the heart to pump the blood into the arterial system. It was captured electronically via an automated record-keeping system. CVP were recorded by experienced anesthesiologists with expertise and qualifications in TEE at five key time points: before surgical incision, start of the preanhepatic phase, start of the anhepatic phase, start of the postanhepatic phase, and after closure of the deep fascial layer of the anterior abdominal wall.
  Low CVP (< 2 mmHg) suggests hypovolemia, dehydration, or blood loss, while normal CVP (2-8 mmHg) indicates balanced fluid status. A high CVP (> 8 mmHg) may indicate fluid overload, right heart failure, pulmonary hypertension, or cardiac tamponade.
Time Frame: From the time patients enter the operating room to leaving the operating room, up to 24 hours.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Measurements
Arm/Group | Liver Transplantation Patients
Number analyzed (Participants) | 58
Number analyzed (Measurements) | 275
mmHg | 11.7 (4.9)

2. Primary Outcome: Correlation of Central Venous Pressure (CVP) and Superior Vena Cava (SVC) Collapsibility Index
Description: The Superior Vena Cava (SVC) Collapsibility Index is used to assess intravascular volume status and fluid responsiveness. The Superior Vena Cava (SVC) collapsibility index was obtained from (Maximum Diameter-Minimum Diameter)/(Maximum Diameter)*100%. Central Venous Pressure (CVP) and SVC were recorded simultaneously by experienced anesthesiologists with expertise and qualifications in TEE at five key time points: before surgical incision, start of the preanhepatic phase, start of the anhepatic phase, start of the postanhepatic phase, and after closure of the deep fascial layer of the anterior abdominal wall.
  The interpretation of the SVC Collapsibility Index is categorized as follows: < 20% indicates low collapsibility, suggesting adequate or high intravascular volume; 20-36% represents an indeterminate zone, requiring additional assessment to determine fluid responsiveness; and > 36% reflects high collapsibility, suggesting hypovolemia or significant fluid deficit.
Time Frame: From the time patients enter the operating room to leaving the operating room, up to 24 hours.
Measure: Mean (Standard Deviation); unit: index
Units Other Than Participants: Measurements
Arm/Group | Liver Transplantation Patients
Number analyzed (Participants) | 58
Number analyzed (Measurements) | 269
index | 26 (11)
Statistical Analysis 1: Comparison: Liver Transplantation Patients; Test type: Superiority; p = 0.944, Repeated measures correlation (rmcorr); correlation coefficient = 0.0005, 98.3% CI 2-sided [-0.161 to 0.170] — The repeated measures correlation coefficient (r_rm) was calculated to assess the association between SVC and CVP. It ranges from -1 to +1, with values closer to +1 indicating that increases in SVC are associated with increases in CVP, and vice versa

3. Primary Outcome: Correlation of Central Venous Pressure (CVP) and Minimum Diameter of Superior Vena Cava (SVC)
Description: The diameter of Superior Vena Cava (normal diameter: 12-22 mm) ) was obtained using transesophageal echocardiography (TEE). Central Venous Pressure (CVP) and SVC were recorded simultaneously by experienced anesthesiologists with expertise and qualifications in TEE at five key time points: before surgical incision, start of the preanhepatic phase, start of the anhepatic phase, start of the postanhepatic phase, and after closure of the deep fascial layer of the anterior abdominal wall.
Time Frame: From the time patients enter the operating room to leaving the operating room, up to 24 hours.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Measurements
Arm/Group | Liver Transplantation Patients
Number analyzed (Participants) | 58
Number analyzed (Measurements) | 269
mm | 12.8 (3.1)
Statistical Analysis 1: Comparison: Liver Transplantation Patients; Test type: Superiority; p < 0.001, Repeated measures correlation (rmcorr); correlation coefficient = 0.27, 98.3% CI 2-sided [0.11 to 0.42] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Correlation of Central Venous Pressure (CVP) and Maximum Diameter of Superior Vena Cava (SVC)
Description: The diameter of the Superior Vena Cava (normal diameter: 12-22 mm) ) was obtained using transesophageal echocardiography (TEE). Central Venous Pressure (CVP) and SVC were recorded simultaneously by experienced anesthesiologists with expertise and qualifications in TEE at five key time points: before surgical incision, start of the preanhepatic phase, start of the anhepatic phase, start of the postanhepatic phase, and after closure of the deep fascial layer of the anterior abdominal wall.
Time Frame: From the time patients enter the operating room to leaving the operating room, up to 24 hours.
Population: maximum Superior Vena Cava (SVC)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Measurements
Arm/Group | Liver Transplantation Patients
Number analyzed (Participants) | 58
Number analyzed (Measurements) | 269
mm | 17.3 (3.2)
Statistical Analysis 1: Comparison: Liver Transplantation Patients; Test type: Superiority; p < 0.001, Repeated measures correlation (rmcorr); correlation coefficient = 0.34, 98.3% CI 2-sided [0.19 to 0.48] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Cardiac Index
Description: The Cardiac Index measures the efficiency of the heart's pumping function (normal range: 2.6 to 4.2 L/min/m2). It was captured electronically via an automated record-keeping system. Cardiac Index was recorded by experienced anesthesiologists with expertise and qualifications in TEE at five key time points: before surgical incision, start of the preanhepatic phase, start of the anhepatic phase, start of the postanhepatic phase, and after closure of the deep fascial layer of the anterior abdominal wall.
Time Frame: From the time patients enter the operating room to leaving the operating room, up to 24 hours.
Measure: Mean (Standard Deviation); unit: L/min/m2
Units Other Than Participants: Measurements
Arm/Group | Liver Transplantation Patients
Number analyzed (Participants) | 58
Number analyzed (Measurements) | 269
L/min/m2 | 4.4 (1.5)

6. Secondary Outcome: Correlation of Cardiac Index (CI) and Superior Vena Cava (SVC) Collapsibility Index
Description: as for outcome 2
Time Frame: From the time patients enter the operating room to leaving the operating room, up to 24 hours.
Measure: Mean (Standard Deviation); unit: index
Units Other Than Participants: Measurements
Arm/Group | Liver Transplantation Patients
Number analyzed (Participants) | 58
Number analyzed (Measurements) | 269
index | 26 (11)
Statistical Analysis 1: Comparison: Liver Transplantation Patients; Test type: Superiority; p = 0.298, Repeated measures correlation (rmcorr); correlation coefficient = 0.07, 98.3% CI 2-sided [-0.10 to 0.24] — The repeated measures correlation coefficient (r_rm) was calculated to assess the association between SVC and CI. It ranges from -1 to +1, with values closer to +1 indicating that increases in SVC are associated with increases in CI, and vice versa

7. Secondary Outcome: Correlation of Cardiac Index (CI) and Minimum Diameter of Superior Vena Cava (SVC)
Description: The diameter of the Superior Vena Cava (normal diameter: 12-22 mm) ) was obtained using transesophageal echocardiography (TEE). Cardiac Index and Superior Vena Cava (SVC) were recorded simultaneously by experienced anesthesiologists with expertise and qualifications in TEE at five key time points: before surgical incision, start of the preanhepatic phase, start of the anhepatic phase, start of the postanhepatic phase, and after closure of the deep fascial layer of the anterior abdominal wall.
Time Frame: From the time patients enter the operating room to leaving the operating room, up to 24 hours.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Measurements
Arm/Group | Liver Transplantation Patients
Number analyzed (Participants) | 58
Number analyzed (Measurements) | 269
mm | 12.8 (3.1)
Statistical Analysis 1: Comparison: Liver Transplantation Patients; Test type: Superiority; p = 0.002, Repeated measures correlation (rmcorr); correlation coefficient = 0.22, 98.3% CI 2-sided [0.05 to 0.37] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Correlation of Cardiac Index (CI) and Maximum Diameter of Superior Vena Cava (SVC)
Description: as for outcome 7
Time Frame: From the time patients enter the operating room to leaving the operating room, up to 24 hours.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Measurements
Arm/Group | Liver Transplantation Patients
Number analyzed (Participants) | 58
Number analyzed (Measurements) | 269
mm | 17.3 (3.2)
Statistical Analysis 1: Comparison: Liver Transplantation Patients; Test type: Superiority; p < 0.001, Repeated measures correlation (rmcorr); correlation coefficient = 0.33, 98.3% CI 2-sided [0.17 to 0.47] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: From the time patients enter the operating room to leaving the operating room, up to 24 hours.
Arm/Group | Liver Transplantation Patients
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT02818218/Prot_SAP_000.pdf